CLINICAL TRIAL: NCT01758809
Title: Pain Control of Thoracoscopic Major Pulmonary Resection: Is Pre-emptive Local Bupivacaine Injection Able to Replace the Intravenous Patient Controlled Analgesia?
Brief Title: Pain Control of Thoracoscopic Major Pulmonary Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Sanghoon Jheon, Chief, Department of Thoracic and Cardiovascular Surgery, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1009-111-015
Record Dates: First submitted 2011-09-28; First posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-12

CONDITIONS: Postoperative Pain
Keywords: Video Assisted Thoracic Surgery; Postoperative Pain; Intravenous Patient Controlled Analgesia; Bupivacaine; Major Pulmonary Resection; Post Pulmonary Resection
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine (Active Comparator)
  Interventions: Procedure: Pre-emptive bupivacaine wound infiltration
- Intravenous Patient Controlled Analgesia (Other): postoperative pain control with intravenous patient controlled analgesia
  Interventions: Procedure: intravenous patient controlled analgesia

INTERVENTIONS:
Procedure: Pre-emptive bupivacaine wound infiltration — Pre-emptive bupivacaine wound infiltration
  Arms: Bupivacaine
Procedure: intravenous patient controlled analgesia — postoperative pain control with intravenous patient controlled analgesia
  Arms: Intravenous Patient Controlled Analgesia

SUMMARY:
The purpose of this study is to evaluate whether pre-emptive local bupivacaine injection is a better alternative pain control modality than the conventional intravenous patient controlled analgesia.

DETAILED DESCRIPTION:
Despite less postoperative pain from Video Assisted Thoracic Surgery (VATS) than thoracotomy, pain is still an important issue in its recovery period. After VATS procedure, intravenous patient controlled analgesia (IV PCA) is being used for pain control. However, the side effects of IV PCA are nausea, vomiting, sleepiness, and urination difficulty which interrupt the early recovery. It is established that pre-emptive local bupivacaine injection is more economical, has almost no side effects, and finally, it is effective for the postoperative 24 hours. The purpose of this study is to evaluate whether pre-emptive local bupivacaine injection is a better alternative pain control modality than the conventional intravenous patient controlled analgesia.

ELIGIBILITY:
Inclusion Criteria:

* patients that are expected to receive VATS segmenectomy or lobectomy regardless of disease entity

Exclusion Criteria:

* not done by VATS anatomical resection
* patient does not agree to the study
* postoperative hospital stay exceeds 7 days due to postoperative complications
* existence of preoperative renal insufficiency (Cr > 1.5)
* OT/PT > 120
* history of Lidocaine hypersensitivity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The change in postoperative pain confirmed by Visual Analogue Pain Scale | Operation day, Postoperative Day 1, 2, 3 and 2 week, 1 month, 2 months

SECONDARY OUTCOMES:
number of participants with adverse events related to fentanyl or bupivacaine drug | 2 months
  nausea, vomiting, sleepiness, urinary difficulty, respiratory depression

CONTACTS AND LOCATIONS:
Overall Officials: Sanghoon Jheon, M.D., Ph.D., Study Chair — Seoul National University Bundang Hospital; Hee Chul Yang, M.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea